CLINICAL TRIAL: NCT05337436
Title: Ionized Magnesium Balance During Hemodialysis Session
Acronym: MAGNESIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0004
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease patient on dialysis (stage 5D); Extracorporeal purification; Ionized magnesium
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients receive conventional dialysis treatment at enrollment: All patients receive conventional dialysis treatment at enrollment
  Interventions: Biological: Lymphatic drainage; Biological: Total and ionized magnesium; Biological: Total and ionized calcium

INTERVENTIONS:
Biological: Lymphatic drainage — Biological determination in plasma:
  Other Names: Biological determination in plasma:
Biological: Total and ionized magnesium — Total and ionized magnesium
Biological: Total and ionized calcium — Total and ionized calcium

SUMMARY:
Aim of this study is to evaluate in a population of chronic kidney disease patients on dialysis (Stage 5D) the balance of total and ionized magnesium according to different types of dialysate used in clinical practice (acetate + Mg 0.50 or 0.75 mM vs citrate + Mg 0.50 ou 0.75 mM)

ELIGIBILITY:
Inclusion criteria:

* Chronic Kidney Disease patient on dialysis (stage 5D) for more than 1 month
* Anuric patient

Exclusion criteria:

* Patient protected by law
* Patient under guardianship ou curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients issued from dialysis units (non profit dialysis centers)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of ionized magnesium levels before and after dialysis session | day 1
  Comparison of ionized magnesium levels before and after dialysis session

SECONDARY OUTCOMES:
Comparison of total magnesium levels before and after dialysis session | day 1
  Comparison of total magnesium levels before and after dialysis session
Comparison of ionized calcium levels before and after dialysis session | day 1
  Comparison of ionized calcium levels before and after dialysis session
Comparison of total calcium levels before and after dialysis session | day 1
  Comparison of total calcium levels before and after dialysis session
Per-dialytic balance of ionized magnesium according to predialysis level | day 1
  Per-dialytic balance of ionized magnesium according to predialysis level
Per-dialytic balance of total magnesium according to predialysis level | day 1
  Per-dialytic balance of total magnesium according to predialysis level
Per-dialytic balance of ionized calcium according to predialysis level | day 1
  Per-dialytic balance of ionized calcium according to predialysis level
Per-dialytic balance of total calcium according to predialysis level | day 1
  Per-dialytic balance of total calcium according to predialysis level

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Study Director — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC